CLINICAL TRIAL: NCT06117254
Title: Evaluating Device-based Rehabilitation for Veterans With Functional Hearing Difficulties: A Randomized Controlled Trial
Brief Title: Hearing Aids for Veterans With Functional Hearing Difficulties
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C4791-R
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Auditory Processing Disorder
Keywords: Auditory Perception; Hearing; Acoustic Stimulation
MeSH Terms: conditions — Auditory Perceptual Disorders | interventions — Hearing Aids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Communication Counseling (Active Comparator): Individuals randomized to this group will receive information on how to improve their ability to hear and communicate including tips on environmental modification and communication repair strategies.
  Interventions: Behavioral: Communication Counseling
- Hearing Aids (Experimental): Individuals randomized to this group will receive communication counseling as well as hearing aids set to provide a low level of amplification.
  Interventions: Behavioral: Communication Counseling; Device: Hearing Aids
- Hearing Aids with Remote Microphones (Experimental): Individuals randomized to this group will receive communication counseling as well as hearing aids set to provide a low level of amplification and remote microphones that can be used in some situations to improve the signal-to-noise ratio.
  Interventions: Behavioral: Communication Counseling; Device: Hearing Aids; Device: Remote Microphones

INTERVENTIONS:
Behavioral: Communication Counseling — Individuals randomized to this group will receive information on how to improve their ability to hear and communicate including general tips on environmental modification and communication repair strategies and personalized tips to help with patient-specific listening difficulties. This is consistent with current audiological standard of care.
Device: Hearing Aids — Hearing aids will be provided with amplification settings programmed specific to each participant's pure-tone hearing thresholds with subsequent adjustments based upon participant preferences. Standard noise cancelation and signal-to-noise ratio improvement strategies will be activated.
  Arms: Hearing Aids; Hearing Aids with Remote Microphones
Device: Remote Microphones — Remote microphone systems will be provided for use with hearing aids.
  Arms: Hearing Aids with Remote Microphones

SUMMARY:
Every year, approximately 100,000 Veterans seek help at VA Audiology clinics for hearing and communication difficulties only to learn that they have normal hearing sensitivity. Unfortunately, there are very few established options to improve hearing and listening for these patients. To address this need, audiologists are increasingly prescribing hearing aids set to provide a small amount of amplification. Patients may benefit from the amplification or from modern hearing aid features such as noise reduction technology and the ability to stream sounds from a desired sound source directly to their ears thus reducing the background noise. This project will help to determine if prescribing hearing aids to patients without hearing loss is, in fact, beneficial and if so, why. It will also help to determine if some patients benefit more from hearing aids than others so that in the future, rehabilitation strategies can be better targeted toward individuals.

DETAILED DESCRIPTION:
At least 10% of Veterans seeking help in VA audiology clinics have clinically normal audiograms, a figure that broadly confirms a recent prevalence study indicating that 33.6% of current active-duty military Service Members are at risk of hearing and communication deficits despite having normal-hearing thresholds. While a considerable amount of research effort over the past 20 years has been devoted to understanding the potential causes for hearing difficulties in patients with normal hearing sensitivity, comparatively little research effort has been devoted to rehabilitation and improvement of function for these patients. This predicament has left audiologists and other medical professionals with very few evidence-based options to provide care for the large segment of help-seeking Veterans struggling with functional hearing difficulties. Currently, audiologic standard of care (SOC) for these patients involves reassurance of normal hearing and providing general communication tips, though evidence suggests that many patients are unsatisfied with this approach and request further testing and rehabilitation options. To help address patient concerns, many VA audiologists are now prescribing hearing aids though there is very little data on whether these devices improve functional outcomes for patients with self-reported hearing difficulties and normal hearing sensitivity. Therefore, the purpose of this study is to compare the efficacy of device-based rehabilitation options with current standard of care for Veterans with self-reported hearing and communication problems, and to identify subgroups in the sample that may benefit differently depending upon patient-specific characteristics and needs. The general hypothesis is that most Veterans with hearing difficulties and normal audiograms will benefit from device-based auditory rehabilitation as reflected by decreases in perceived hearing handicap. However, the amount of benefit will vary according to patient-specific characteristics including auditory, psychological and cognitive factors in combination with the type and severity of auditory dysfunction experienced by the patient.

All study participants will be Veterans with normal to near-normal pure-tone sensitivity but with moderate to severe perceived hearing handicap who are interested in seeking professional help. Participants will be interviewed to gather data regarding their hearing difficulties, including the context and impacts of difficulties as well as goals for auditory rehabilitation. Next, participants will undergo assessments of peripheral and central auditory system function including electrophysiological and behavioral measures and cognitive and psychological status assessed using established NIH Toolbox® measures. Participant medical charts will be reviewed to gather data on comorbid conditions and previous exposures known to be risk factors for developing auditory processing difficulties. These data will be compiled to provide an estimate of the distribution of characteristics likely to impact auditory function and response to intervention among Veterans seeking help for functional hearing difficulties. Participants will then be randomized into one of following three intervention arms: 1. SOC, 2. SOC + hearing aids, or 3. SOC + hearing aids with remote microphone. Outcomes will be measured at two- and six-months post-intervention. The primary outcome measure is the Hearing Handicap Inventory for Adults. Secondary outcome measures are aimed at identifying the underlying mechanisms and potential mediators that influence whether and how participants receive benefit from hearing devices. These will include measures of speech understanding in quiet and noise, objective and subjective listening effort, electrophysiological measures of neural responses to sound, and interviews to learn more about participants' perceptions of the intervention. Interaction effects will be estimated between treatment arm and patient characteristics to identify key moderating factors that influence the degree and direction of benefit associated with different treatment strategies. This information can then be used to inform both clinical decision making for individual patients and the design of future intervention studies.

ELIGIBILITY:
Inclusion Criteria:

* Veteran eligible for VA Healthcare
* Ability to travel to VA Portland Medical Center for repeated visits
* Pure-tone thresholds of no more than 30 dB HL at frequencies between 500 and 3000 Hz, and no more than 40 dB HL at 4000 Hz
* HHIA scores of 24 or greater indicating moderate to significant perceived hearing handicap

Exclusion Criteria:

* Conductive hearing loss or other significant otologic problems
* Non-native English speakers
* Inability to perform experimental tasks
* Pure-tone interaural threshold asymmetries greater than 15 dB between 250 and 4000 Hz

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2025-03-09 (Actual); Primary Completion 2027-10-29 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Hearing Handicap Inventory for Adults (HHIA) score | Baseline and 2- and 6-months post randomization
  The HHIA is a self-report measure of the impact of hearing difficulties on daily life and functioning, including social and emotional affects. It is comprised of 25 questions with total scores from 0 to 100. Higher scores indicate greater levels of perceived hearing handicap.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa A Papesh, PhD, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No